CLINICAL TRIAL: NCT07176416
Title: Assessment of Effective Phaco Time and Endothelial Cell Loss When Using a Novel Dual Mode Phacoemulsification System
Brief Title: Effective Phaco Time and Endothelial Cell Loss When Using Veritas
Status: Recruiting | Type: Observational
Sponsor: Aloha Vision Consultants (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: CY-25-01
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Veritas Vision System — Veritas Vision System

SUMMARY:
This study is a single center, prospective study of cumulative dissipated energy and endothelial cells loss per phacoemulsification procedure after successful cataract surgery. Subjects will be assessed 3 months postoperatively at a single visit. Clinical evaluations will include central corneal thickness, specular microscopy, as well as measurement of visual acuities at distance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing age-related cataract surgery.
* Planned use of the Catalys Precision Laser System.
* Planned implantation of TECNIS intraocular lenses (IOLs).

Exclusion Criteria:

• Moderate-severe any disease state (deemed by the surgeon) that could increase risk of complicated cataract surgery (ie, pseudoexfoliation syndrome, zonular dehiscence, history of eye trauma, and prior refractive surgery).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible test subjects will be adults who are candidates for age-related cataract surgery with IOL implantation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Effective phaco time per phacoemulsification procedure | Surgery (Day 0)

SECONDARY OUTCOMES:
Endothelial cell loss | 1 monthspostoperatively
Total case time | Surgery (Day 0)
  total case time per procedure
Total phaco time | Surgery (Day 0)
  total phaco time per procedure
Total volume used | Surgery (Day 0)
  Total volume used per procedure

CONTACTS AND LOCATIONS:
Overall Officials: Carlton Yuen, MD, Principal Investigator — Aloha Vision Consultants
Locations (1):
- Aloha Vision Consultants, ‘Aiea, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No